CLINICAL TRIAL: NCT01684982
Title: Randomized Comparison of Everolimus Eluting Stents and Sirolimus Eluting Stent in Patients With ST Elevation Myocardial Infarction (STEMI) (RaCES-MI Trial)
Brief Title: Everolimus Stent in Myocardial Infarction
Acronym: RaCES-MI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: San Giuseppe Moscati Hospital (Other)
Responsible Party: Principal Investigator, Emilio Di Lorenzo MD PhD, Chief Interventional Cardiology, San Giuseppe Moscati Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DiLOR_2012
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Acute Myocardial Infarction
Keywords: Primary PCI; Drug Eluting Stent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- everolimus eluting stent (Experimental): second generation drug eluting stent
  Interventions: Device: everolimus eluting stent
- sirolimus eluting stent (Active Comparator): first generation drug eluting stent
  Interventions: Device: sirolimus eluting stent

INTERVENTIONS:
Device: everolimus eluting stent — experimental arm of a comparison between drug eluting stents
  Other Names: XIENCE V Abbott Vascular
  Arms: everolimus eluting stent
Device: sirolimus eluting stent — control arm of a comparison between drug eluting stents
  Other Names: CYPHER Johnson & Johnson
  Arms: sirolimus eluting stent

SUMMARY:
Randomized trial to test the efficacy and safety of newer Drug Eluting Stent generation in patient with acute myocardial infarction treated with primary percutaneous coronary intervention (PCI)

DETAILED DESCRIPTION:
The efficacy and safety of drug-eluting stents (DES) in the treatment of coronary artery disease is well established. It is well known that Drug Eluting Stent (DES) have dramatically decreased Restenosis rates for both on-label and off-label indications. However, the concern for increased (late) stent thrombosis is still present DES implantation in patient with acute myocardial infarction is still controversial because acute coronary lesion presents the highest possible thrombotic burden Newer DES with new antiproliferative drugs and more biocompatible polymers have shown a significant reduction of (late) stent thrombosis in patients in stable condition.

Aim of the study was to asses the long term efficacy and safety on second generation everolimus eluting stent compared with first generation sirolimus eluting stent

ELIGIBILITY:
Inclusion Criteria:

* All ST segment elevation myocardial infarction (STEMI) patients eligible for primary PCI

Exclusion Criteria:

1. Contraindication to dual antiplatelet therapy for 12 months
2. Known allergy to sirolimus or everolimus
3. Major surgical procedure planned within 1 month.
4. History, symptoms, or findings suggestive of aortic dissection.
5. Participation in other trials
6. Pregnancy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2007-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
cardiac death, reinfarction and Target Vessel Revascularization (TVR) | 36 MONTHS
  Any death of cardiac origin, any myocardial infarction and any new revascularization of the infarct related artery

SECONDARY OUTCOMES:
cardiac death, reinfarction, Target Vessel Revascularization (TVR) and definite/probable stent thrombosis | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: EMILIO DI LORENZO, MD PHD, Principal Investigator — AO MOSCATI AVELLINO ITALY; ROSARIO SAURO, MD, Study Director — AO MOSCATI AVELLINO ITALY
Locations (1):
- Division of Cardiology AO Moscati, Avellino, Italy

REFERENCES:
- [Background] De Luca G, Dirksen MT, Spaulding C, Kelbaek H, Schalij M, Thuesen L, van der Hoeven B, Vink MA, Kaiser C, Musto C, Chechi T, Spaziani G, Diaz de la Llera LS, Pasceri V, Di Lorenzo E, Violini R, Cortese G, Suryapranata H, Stone GW; Drug-Eluting Stent in Primary Angioplasty (DESERT) Cooperation. Drug-eluting vs bare-metal stents in primary angioplasty: a pooled patient-level meta-analysis of randomized trials. Arch Intern Med. 2012 Apr 23;172(8):611-21; discussion 621-2. doi: 10.1001/archinternmed.2012.758. PMID 22529227
- [Background] Di Lorenzo E, Carbone G, Sauro L, Casafina A, Capasso M, Sauro R. Bare-metal stents versus drug-eluting stents for primary angioplasty: long-term outcome. Curr Cardiol Rep. 2011 Oct;13(5):459-64. doi: 10.1007/s11886-011-0207-0. PMID 21792636
- [Background] Dibra A, Tiroch K, Schulz S, Kelbaek H, Spaulding C, Laarman GJ, Valgimigli M, Di Lorenzo E, Kaiser C, Tierala I, Mehilli J, Campo G, Thuesen L, Vink MA, Schalij MJ, Violini R, Schomig A, Kastrati A. Drug-eluting stents in acute myocardial infarction: updated meta-analysis of randomized trials. Clin Res Cardiol. 2010 Jun;99(6):345-57. doi: 10.1007/s00392-010-0133-y. Epub 2010 Mar 11. PMID 20221617
- [Background] Di Lorenzo E, Sauro R, Varricchio A, Capasso M, Lanzillo T, Manganelli F, Mariello C, Siano F, Pagliuca MR, Stanco G, Rosato G, De Luca G. Benefits of drug-eluting stents as compared to bare metal stent in ST-segment elevation myocardial infarction: four year results of the PaclitAxel or Sirolimus-Eluting stent vs bare metal stent in primary angiOplasty (PASEO) randomized trial. Am Heart J. 2009 Oct;158(4):e43-50. doi: 10.1016/j.ahj.2009.03.016. PMID 19781402
- [Background] Hofma SH, Brouwer J, Velders MA, van't Hof AW, Smits PC, Quere M, de Vries CJ, van Boven AJ. Second-generation everolimus-eluting stents versus first-generation sirolimus-eluting stents in acute myocardial infarction. 1-year results of the randomized XAMI (XienceV Stent vs. Cypher Stent in Primary PCI for Acute Myocardial Infarction) trial. J Am Coll Cardiol. 2012 Jul 31;60(5):381-7. doi: 10.1016/j.jacc.2012.01.073. PMID 22835668
- [Background] Sabate M, Cequier A, Iniguez A, Serra A, Hernandez-Antolin R, Mainar V, Valgimigli M, Tespili M, den Heijer P, Bethencourt A, Vazquez N, Gomez-Hospital JA, Baz JA, Martin-Yuste V, van Geuns RJ, Alfonso F, Bordes P, Tebaldi M, Masotti M, Silvestro A, Backx B, Brugaletta S, van Es GA, Serruys PW. Everolimus-eluting stent versus bare-metal stent in ST-segment elevation myocardial infarction (EXAMINATION): 1 year results of a randomised controlled trial. Lancet. 2012 Oct 27;380(9852):1482-90. doi: 10.1016/S0140-6736(12)61223-9. Epub 2012 Sep 3. PMID 22951305
- [Derived] Di Lorenzo E, Sauro R, Varricchio A, Capasso M, Lanzillo T, Manganelli F, Carbone G, Lanni F, Pagliuca MR, Stanco G, Rosato G, Suryapranata H, De Luca G. Randomized comparison of everolimus-eluting stents and sirolimus-eluting stents in patients with ST elevation myocardial infarction: RACES-MI trial. JACC Cardiovasc Interv. 2014 Aug;7(8):849-56. doi: 10.1016/j.jcin.2014.02.016. PMID 25147029